CLINICAL TRIAL: NCT03467854
Title: Pharmacokinetics (PK) of Piperacillin/Tazobactam in Adults Undergoing Extracorporeal Membrane Oxygenation (ECMO)
Brief Title: PK of Piperacillin/Tazobactam in Adults Undergoing ECMO
Status: Terminated | Type: Observational
Why Stopped: Lack or eligible patients.
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Darryl Abrams, Professor of Medicine, Columbia University
Other Study IDs: AAAR7200
Record Dates: First submitted 2018-03-10; First posted 2018-03-16 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Acute Respiratory Failure With Hypoxia
Keywords: ECMO; Antimicrobials

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Four blood samples will be obtained after the first dose of piperacillin/tazobactam: one sample before the second dose, 30-minutes, 2-hours, and 6-hours into the infusion. An additional four blood samples will be drawn on day 2 at the same time points.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- VV ECMO: Patients 18 years of age or older, initiated on veno-venous (VV) ECMO for acute respiratory distress syndrome, and receiving piperacillin/tazobactam.Four blood samples will be obtained after the first dose of piperacillin/tazobactam: one sample before the second dose, 30-minutes, 2-hours, and 6-hours into the infusion. An additional four blood samples will be drawn on day 2 at the same time points.

SUMMARY:
This study is designed to provide preliminary data to determine if concentrations of piperacillin/tazobactam change in patients with severe respiratory failure receiving extracorporeal membrane oxygenation (ECMO). The investigators hypothesize that patients will have significant changes in concentration measurements, specifically an increased clearance rate and increased volume of distribution, during ECMO as compared to critically ill patients.

DETAILED DESCRIPTION:
In a healthy patient, the lungs provide oxygen to the blood and remove carbon dioxide. However, in patients with severe lung failure, blood may not adequately be delivered to the lungs, or the lungs may not adequately supply blood with oxygen. In this case, patients may require assistance from a machine to help provide this oxygen. Extracorporeal membrane oxygenation (ECMO) is a device that acts as an artificial lung, allowing the patient to recover from their illness. Patients receiving support from ECMO are often put in a medically induced coma while their lungs heal. Certain drugs may stick to the internal surfaces of the machine; therefore leading to decreased concentrations. Patients receiving ECMO often require antimicrobials to treat severe infections. However, little data exist concerning the likely changes in drug concentrations from drug circuit interactions in adult patients receiving ECMO.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Initiated on VV ECMO for acute respiratory distress syndrome
* Receiving piperacillin/tazobactam

Exclusion Criteria:

* Pregnancy
* Massive blood transfusion (10 units or more of of PRBC) within a 24-hour period
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients receiving VV ECMO for acute respiratory distress syndrome will be assessed for inclusion into the study.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Change in clearance rate | Up to 2 days after the first dose of piperacillin/tazobactam
Change in volume of distribution | Up to 2 days after the first dose of piperacillin/tazobactam

CONTACTS AND LOCATIONS:
Overall Officials: Darryl Abrams, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center / NewYork-Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No